CLINICAL TRIAL: NCT00885339
Title: Evaluation of the PillCam Colon Capsule Endoscopy Preparation and Procedure
Brief Title: Evaluation of the PillCam™ Colon Capsule Endoscopy (PCCE) Preparation and Procedure
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-109
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2010-03

CONDITIONS: Colonic Diseases
Keywords: Colonic Diseases
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases.

SUMMARY:
The purpose of this study is to compare two preparation and procedure in order to develop the most optimal capsule procedure in regards to colon cleansing level and capsule excretion rate.

DETAILED DESCRIPTION:
The evaluation of subjects with suspected colonic disease includes endoscopic imaging by colonoscopy and radiologic imaging such as air-contrast barium enema, or CT colonography. The PillCam platform offers an alternative approach for endoscopic visualization of the colon using capsule endoscopy, an ingestible device which contains imagers, light sources, a power source and a RF transmitter. Advantages of the PillCam platform include the elimination of the need for sedation, the minimally invasive, painless nature of the exam, and the ability to pursue normal daily activities immediately following the procedure . Furthermore, compared to standard colonoscopy, the PillCam platform may be more readily accepted by the subjects, thereby improving subjects' willingness to undergo a diagnostic evaluation of the colon and comply with colorectal cancer screening recommendations.

The PillCam™ SB capsule (formerly M2A® Capsule) that was FDA-approved in August 2001 for small bowel evaluation has been ingested to date by more than 500,000 people worldwide and is well accepted by patients and physicians as well as the processional societies. However, adequate visualization of the colon cannot be achieved with the standard PillCam™ SB capsule because of the anatomical and physiological properties of the colon which are significantly different than the small bowel. Moreover, other issues that limit the evaluation of the colonic mucosa by the standard PillCam™ SB procedure include an unsatisfactory level of colon cleanliness and slow progression of the PillCam™ SB capsule through the colon during the desired examination time. Therefore, the development and introduction of a specially designed, customized colon capsule combined with a dedicated capsule colonoscopy procedure protocol will allow for more efficient evaluation of the colonic mucosa. This is expected to improve the capability of the PillCam platform to detect colonic pathologies and to serve as a diagnostic and screening tool for colonic disease. Further details of the PillCam™ Colon Capsule Endoscope (PCCE) can be found in the device description section.

This is a pilot study that is designed to compare the levels of cleanliness and visualization of colon achieved by colon capsule endoscopy when using two different regimens for preparation of the colon. Furthermore, capsule colonoscopy and colonoscopy procedures will be compared in regards to the level of colon cleanliness and detection of lesions in the colon. The study will be conducted in 2 phases: pilot phase in which the optimal procedure will be determined following a comparison of the two procedures. The second phase will be a validation of the proposed procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between the ages of 18-75 years.
* Subject is referred for colonoscopy as clinically indicated for any reason. This may include, but not limited to, the investigation of any of the following conditions: rectal bleeding, melena, positive stool testing for occult blood, recent change of bowel habits, screening for colorectal cancer, ulcerative colitis, colonic findings on an imaging study)

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

* Subject has dysphagia or any swallowing disorder
* Subject has Congestive heart failure
* Subject has high degree of renal insufficiency
* Subject has had prior abdominal surgery of the gastrointestinal tract other than uncomplicated procedures that would be unlikely to lead to bowel obstruction based on the clinical judgment of the investigator
* Subject has a cardiac pacemaker or other implanted electromedical device.
* Subject has any allergy or other known contraindication to the medications used in the study
* Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
* Subject with any condition believed to have an increased risk for capsule retention such as Crohn's disease, intestinal tumors, radiation enteritis, or NSAID enteropathy,
* Subject has any condition, which precludes compliance with study and/or device instructions.
* Women who are either pregnant or nursing at the time of screening, who intend to be during the study period, or are of child-bearing potential and do not practice medically acceptable methods of contraception.
* Subject suffers from life threatening conditions
* Subject currently participating in another clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are indicated for colonoscopy, who are suspected or known to suffer from colonic diseases
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Colon cleansing level score | within 7 days
Number of colon capsules excreted over time | within 7 days

SECONDARY OUTCOMES:
Accuracy parameters of PCCE, compared to colonoscopy. | within 7 days
Number, type and severity of adverse events | within 7 days
Patient subjective assessment questionnaires | within 7 days
Physician assessment questionnaire | within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Guido Costamagna, Prof. Dr., Principal Investigator — Catholic University of the Sacred Heart
Locations (4):
- Italy (4):
  - Centro Ricerca e Formazione ad Alta Tecnologia nelle Scienze Bomediche, Campobasso
  - Humanitas Istituto Clinico, Milan
  - Ospedale Maggiore - Policlinico, Milan
  - Universita Cattolica del Sacro Cuore, Roma